CLINICAL TRIAL: NCT03847610
Title: Microneedle Sensing of Beta-lactam Antibiotic Concentrations in Human Interstitial Fluid
Brief Title: Minimally Invasive Sensing of Beta-lactam Antibiotics
Acronym: MISBL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 17IC4051; 236047 (Other: IRAS); 18/LO/0054 (Other: London-Harrow REC)
Record Dates: First submitted 2019-02-07; First posted 2019-02-20 (Actual); Results first posted 2020-12-29 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Penicillin V; Penicillins; Proof of Concept Study; Clinical Trial, Phase I; Microneedle array
MeSH Terms: interventions — Penicillin V

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy volunteer (Experimental)
  Interventions: Drug: Phenoxymethyl Penicillin; Device: Microneedle array

INTERVENTIONS:
Drug: Phenoxymethyl Penicillin — Phenoxymethylpenicillin tablets, 500mg every six hours for six doses, starting the day before study
Device: Microneedle array — The microneedle biosensor will be sited peripherally (on the non-dominant arm) for the duration of the study. It will then be removed.

SUMMARY:
This study is an in-house feasibility study of a microneedle biosensor developed within Imperial College London.

DETAILED DESCRIPTION:
Outline of the study:

This study will comprise the recruitment of 10-15 healthy volunteers. They will be recruited to test the microneedle biosensors and undergo rich plasma sampling with or without tissue microdialysis to calibrate the microneedle biosensor and evaluate its accuracy against current gold standards (i.e. plasma drug concentration and tissue microdialysis). This study will take place at the Imperial Clinical Research Facility (CRF).

Patient identification:

Healthy volunteers will be recruited from a healthy volunteer database held within Imperial College London and via identification of participants within the College. An initial advertisement e-mail will be sent and individuals responding will then followed up by telephone and invited to attend a screening visit at the Imperial CRF. They will be sent the participant information leaflet in advance of this meeting to give them time to consider the information. At this visit a member of the research team will go through the study procedure and answer any questions that the participant has.

Consent procedure:

Healthy volunteers who wish to participate in the study after considering the participant information leaflet will be consented by a trained researcher who will complete the eligibility screening for inclusion into the study.

Study Methodology:

10-15 healthy volunteers will be invited to participate in an exploratory study of the sensor device. On their screening visit routine blood tests will be performed to ensure that the participant is not anaemic and has no evidence of current infection. Before the study day the participant will be required to take 5 doses of oral penicillin to ensure that they are at steady state and to allow for stabilization of tissue distribution. Four of these doses will be taken at 6-hour intervals on the day before they attend the Imperial CRF. The final dose will be taken on the morning that they attend.

On arrival at the study centre the participant will have a microneedle biosensor sited for up to 12 hours whilst receiving antimicrobial therapy. The sensor will be sited peripherally (on an arm or leg). In a small number of cases the sensor may be sited centrally on the torso. These sensors are connected to potentiostat devices that records data, which can then be downloaded onto a computer for analysis.

Following arrival on the study day and placing of the sensor devices, a cannula will be sited for phlebotomy and a baseline beta-lactam antibiotic concentration will be taken. A microdialysis fibre will also be inserted peripherally into tissue close to the microneedle device to allow gold standard analysis of tissue antibiotic concentration. The participant will then undergo rich plasma drug sampling with up to 15 blood tests taken over a 6-12 hour period.

Each blood test will involve the collection of 3mL extra blood (<1 teaspoons) via a cannula which will be cited on commencement of the study. Microdialysis may be performed in all participants who consent to this as a gold standard for determining tissue drug concentrations. If they do not consent for this, the study will be able to continue without microdialysis being performed. Participants will also be required to complete a visual analogue scale every hour testing their level of discomfort due to the microneedle sensor device and a member of the research team will document any redness or skin changes around the site of the device. A further dose of penicillin will be given approximately 6 hours into the study.

Time points for the blood sampling are planned to initially be taken at (0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240, 360, 480, 600, 720 minutes). However, following initial pharmacokinetic (PK) analysis a D-optimal design will be employed using Pmetrics and BestDose PK software to determine the optimal time points for blood PK analysis. This will be performed by a trained member of the research team.

Clinically relevant data including demographic, co-morbidity, and medication data will be collected by members of the research team from the participant.

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 years old
* Healthy with no evidence of active infection
* Previously received penicillin with no adverse effects

Exclusion Criteria:

* High risk of skin soft tissue infection or local skin and soft tissue infection near sensor site
* Previous history of allergies to adhesive strips or active dermatitis
* Penicillin allergy or previous adverse event whilst receiving penicillin
* Anaemia on screening bloods (defined as haemoglobin <13 g/dL in males and <12 g/dL in females)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison H Holmes, MD MPH MBBS, Principal Investigator — Health Protection Research Unit in HCAI & AMR
Locations (1):
- NIHR Imperial CRF, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rawson TM, Gowers SAN, Freeman DME, Wilson RC, Sharma S, Gilchrist M, MacGowan A, Lovering A, Bayliss M, Kyriakides M, Georgiou P, Cass AEG, O'Hare D, Holmes AH. Microneedle biosensors for real-time, minimally invasive drug monitoring of phenoxymethylpenicillin: a first-in-human evaluation in healthy volunteers. Lancet Digit Health. 2019 Nov;1(7):e335-e343. doi: 10.1016/S2589-7500(19)30131-1. Epub 2019 Sep 30. PMID 33323208

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One volunteer withdrew consent to undergo microdialysis on the study day and was withdrawn from the analysis. The participant did not cite a reason for declining microdialysis catheter insertion. Therefore, ten volunteers were included in the study.
Period: Overall Study
Arm/Group | Healthy Volunteer
Started | 11
Completed | 10
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Volunteer
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 10
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24 (3)
Creatinine clearance [Mean (Standard Deviation); unit: mL/min] | 114 (29)
Height [Mean (Standard Deviation); unit: cm] | 174 (11)
Weight [Mean (Standard Deviation); unit: kg] | 74 (15)

OUTCOME MEASURES:

1. Primary Outcome: Assessment of the Biosensors Ability to Track Phenoxymethylpenicillin Concentrations Compared to Observations Made by Microdialysis and Blood Sampling
Description: Bland-Altman plot to describe agreement between interstitial phenoxymethylpenicillin concentrations and microneedle data (mean difference between microneedle and microdialysis measurements)
Time Frame: Up to 12 hours
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Healthy Volunteer
Number analyzed (Participants) | 10
mg/L | -0.16 [-1.3 to 0.82]

ADVERSE EVENTS:
Time Frame: Study day -1, and on the study day for each participant
Arm/Group | Healthy Volunteer
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/10/NCT03847610/Prot_000.pdf